CLINICAL TRIAL: NCT04103424
Title: Mitochondrial Remodeling After Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon State University (Other)
Responsible Party: Principal Investigator, Sean Newsom, Assistant Professor, Oregon State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-2019-0124
Record Dates: First submitted 2019-08-23; First posted 2019-09-25 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Overweight and Obesity; Insulin Resistance; Metabolic Disease; Mitochondrial Metabolism; Sedentary Lifestyle
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Metabolic Diseases; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be asked to complete 2 screening visits to determine eligibility. If participants remain eligible, they will be asked to complete 2 metabolic study visits, 1 before and 1 after 2 weeks of supervised exercise training on a stationary bike.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-training Metabolic Study Visit (No Intervention): Participants will first complete a pre-training metabolic study visit.
- Post-training Metabolic Study Visit (Experimental): Participants will complete a second, identical metabolic study visit following 2-weeks of exercise training.
  Interventions: Behavioral: Short-term Exercise Training

INTERVENTIONS:
Behavioral: Short-term Exercise Training — Participants will perform 2-weeks of supervised exercise training on a stationary bike.
  Arms: Post-training Metabolic Study Visit

SUMMARY:
Regulation of mitochondrial health in overweight and obese individuals may be impaired. The purpose of this study is to identify impairments in regulation of mitochondrial health within skeletal muscle and to determine if short-term exercise training (2-weeks) can reverse such impairments. The investigator's hypothesis is that pathways that serve to degrade poorly functioning mitochondria in overweight and obese individuals are down-regulated, but that short-term exercise training can restore these pathways to improve skeletal muscle mitochondrial function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* Body mass index (BMI) 18-45 kg/m2
* Sedentary (<1 hour of planned exercise per week)

Exclusion Criteria:

* Regular exercise (>1 hour of planned exercise per week)
* Smoking, tobacco or nicotine use within the last 1-year
* Fasting glucose >126mg/dL
* Hypertension (systolic pressure >140 mmHg or diastolic pressure >90 mmHg)
* Chronic metabolic or cardiovascular health conditions
* Pregnant, nursing, irregular menses or post-menopausal
* Lidocaine allergy
* Certain medications
* Physical limitations that prevent safe or successful exercise completion
* Diminished capacity for consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
Change in skeletal muscle mitochondrial protein degradation peptide products | After 2-weeks of exercise training compared with before training.
  Skeletal muscle mitochondrial protein degradation peptide products after 2-weeks of exercise training compared with before training.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Newsom, PhD, Principal Investigator — Oregon State University; Matthew Robinson, PhD, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No